CLINICAL TRIAL: NCT06562231
Title: Development of Isthmocele Symptom Severity and Quality of Life Questionnaire
Brief Title: Development of Isthmocele Symptom Severity and Quality of Life Scale
Status: Recruiting | Type: Observational
Sponsor: Hilal Yuvacı (Other)
Responsible Party: Sponsor-Investigator, Hilal Yuvacı, Obstetrics and Gynecology, Sakarya University
Organization: Sakarya University (Other)
Other Study IDs: isthmocele and quality of life
Record Dates: First submitted 2022-12-20; First posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Quality of Life
Keywords: isthmocele; quality of life; questionnaire; abnormal uterine bleeding
MeSH Terms: conditions — Metrorrhagia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- questionnaire group: The patient will fill out the questionnaire form with the diagnosis of isthmocele.
  Interventions: Other: quality of life scale

INTERVENTIONS:
Other: quality of life scale — This study will be conducted on women diagnosed with symptomatic isthmocele after cesarean section. Researchers will prepare scale questions, and the survey questions will be developed after obtaining an expert opinion from 20 experts to be evaluated by psychiatry, obstetrics, and public health experts. The patient will fill out the questionnaire form with the diagnosis of isthmocele. Oral and written consent will be obtained from the patients.

SUMMARY:
Isthmocele, also known as cesarean scar defect (CSD), is the disruption of the integrity of the myometrium in the cesarean section incision and the indentation of the opening in the myometrium towards the visceral peritoneum. Residual menstrual blood accumulating in the isthmocele sac can cause chronic endometritis, anormal uterine bleeding, infertility and chronic pelvic pain.

There is currently no quality of life scale that assesses isthmocele symptoms. A scale is needed to determine the positive effect on the patient's quality of life after the surgeries are performed. This study it is aimed to develop a scale that evaluates the severity of isthmocele symptoms and the impact on quality of life due to isthmocele.

DETAILED DESCRIPTION:
Patients with isthmocele symptoms three months after cesarean delivery will be included in the study.The study will not include findings that may be confused with isthmocele symptoms, such as uterine fibroids and endometrial polyps. Patients with acute vaginitis and pelvic inflammatory disease will not be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with isthmocele symptoms three months after cesarean delivery will be included in the study.

Exclusion Criteria:

* The study will not include findings that may be confused with isthmocele symptoms, such as uterine fibroids and endometrial polyps.
* Patients with acute vaginitis and pelvic inflammatory disease will not be included in the study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: This study will be conducted on women diagnosed with symptomatic isthmocele after cesarean section.
Sampling Method: Probability Sample
Enrollment: 330 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Development of isthmocele symptom severity and quality of life scale | 3 year
  In the literature review, there is currently no quality of life scale for isthmocele symptoms. There is a need for a scale to detect changes in patients' quality of life after surgery due to isthmocele.This study aimed to create a questionnaire that can be administered immediately before surgery and six weeks after surgery to assess the severity of isthmocele symptoms and the impact of isthmocele on quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Hilal Uslu Yuvacı, Principal Investigator — Sakarya University School of Medicine
Locations (1):
- Sakarya University School of Medicine, Sakarya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2023-01-01): https://cdn.clinicaltrials.gov/large-docs/31/NCT06562231/Prot_000.pdf